CLINICAL TRIAL: NCT02978716
Title: Phase 2 Study of the Safety, Efficacy, and Pharmacokinetics of G1T28 in Patients With Metastatic Triple Negative Breast Cancer Receiving Gemcitabine and Carboplatin Chemotherapy
Brief Title: Trilaciclib (G1T28), a CDK 4/6 Inhibitor, in Combination With Gemcitabine and Carboplatin in Metastatic Triple Negative Breast Cancer (mTNBC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary Analysis and survival follow up completed per protocol. Not stopped due to safety concerns
Sponsor: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G1T28-04; 2016-004466-26 (EudraCT Number)
Record Dates: First submitted 2016-11-18; First posted 2016-12-01 (Estimated); Results first posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-02

CONDITIONS: Triple-Negative Breast Neoplasms; Breast Neoplasm; Breast Cancer; Triple-Negative Breast Cancer
Keywords: Breast Cancer; CDK 4/6 Inhibitor; Triple Negative Breast Cancer; Metastatic
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Neoplasm Metastasis | interventions — trilaciclib; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Gemcitabine/Carboplatin (Days 1 and 8) (Experimental): Participants received Intravenous (IV) infusion of standard GC chemotherapy (gemcitabine 1000 milligrams per meter square [mg/m^2] and carboplatin area under the curve [AUC] 2) on Days 1 and 8 of 21-day cycle. The carboplatin dose was calculated using the Calvert formula, with a target AUC 2 (maximum 300 mg).
  Interventions: Drug: Gemcitabine; Drug: Carboplatin
- Group 2: Trilaciclib + Gemcitabine/ Carboplatin (Days 1 and 8) (Experimental): Participants received IV infusion of trilaciclib 240 mg/m^2 plus GC chemotherapy (gemcitabine 1000 mg/m^2 and carboplatin AUC 2) IV infusion on Days 1 and 8 of 21-day cycle. Trilaciclib was administered prior to chemotherapy.
  Interventions: Drug: Trilaciclib; Drug: Gemcitabine; Drug: Carboplatin
- Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9) (Experimental): Participants received IV infusion of trilaciclib 240 mg/m^2 on Days 1, 2, 8, and 9 plus GC chemotherapy (gemcitabine 1000 mg/m^2 and carboplatin AUC 2) IV infusion on Day 2 and 9 of 21-day Cycle. Trilaciclib was administered prior to chemotherapy.
  Interventions: Drug: Trilaciclib; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Trilaciclib — G1T28
  Other Names: G1T28; CDK 4/6 Inhibitor
  Arms: Group 2: Trilaciclib + Gemcitabine/ Carboplatin (Days 1 and 8); Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Drug: Gemcitabine — Gemcitabine
Drug: Carboplatin — Carboplatin

SUMMARY:
This was a study to investigate the potential clinical benefit of trilaciclib (G1T28) in preserving the bone marrow and the immune system, and enhancing chemotherapy antitumor efficacy when administered prior to carboplatin and gemcitabine (GC therapy) for participants with metastatic triple negative breast cancer.

The study was an open-label and 102 participants were randomly assigned (1:1:1 fashion) to 1 of the 3 following treatment groups:

* Group 1: GC therapy (Days 1 and 8 of 21-day cycles) only (n=34)
* Group 2: GC therapy (Days 1 and 8) plus trilaciclib (G1T28) on Days 1 and 8 of 21-day cycles (n=33)
* Group 3: GC therapy (Days 2 and 9) plus trilaciclib (G1T28) on Days 1, 2, 8, and 9 of 21-day cycles (n=35)

The study included 3 study phases: Screening Phase, Treatment Phase, and Survival Follow-up Phase. The Treatment Phase begins on the day of first dose with study treatment and completes at the Post-Treatment Visit.

DETAILED DESCRIPTION:
The posted results represent the final results of Study G1T28-04, a Phase 2 study of the safety, efficacy and pharmacokinetics of trilaciclib (G1T28) in patients with locally recurrent/metastatic triple negative breast cancer receiving gemcitabine and carboplatin chemotherapy.

The final myelopreservation efficacy results are reported from database lock 1 ([DBL1], data cut-off [DCO] date of 30 July 2018). Final anti-tumor efficacy (ORR, PFS), and final summary exposure and safety data are reported from database lock 2 ([DBL2], DCO 28 June 2019) which occurred to support filing of the trilaciclib New Drug Application (NDA). Final overall survival (OS) data are reported from the final database lock which occurred on 17 July 2020 (with a last patient last visit date of 28 February 2020).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of hormone receptor (HR)-negative, human epidermal growth factor receptor 2 (HER2)-negative (locally recurrent or metastatic TNBC) breast cancer
* Available TNBC diagnostic tumor tissue (archived tissue allowed)
* Evaluable disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Adequate organ function
* Predicted life expectancy of 3 or more months

Exclusion Criteria:

* More than 2 prior chemotherapy regimens for locally recurrent or metastatic TNBC. If > 12 months have elapsed between the date of last adjuvant/neoadjuvant chemotherapy administration and first documented local or distant disease recurrence the therapy will not be considered a line of therapy in the locally recurrent or metastatic TNBC setting.
* CNS metastases or leptomeningeal disease requiring immediate treatment with radiation therapy or steroids.
* Investigational drug within 30 days of first trilaciclib (G1T28) dose
* Concurrent radiotherapy, radiotherapy within 14 days of first trilaciclib (G1T28) dose
* Cytotoxic chemotherapy within 3 weeks of first trilaciclib (G1T28) dose
* Prior hematopoietic stem cell or bone marrow transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Contact, Study Director — G1 Therapeutics, Inc.
Locations (54):
- United States (35):
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Disney Family Cancer Center, Burbank, California
  - Sharp Clinical Oncology, San Diego, California
  - Innovative Clinical Research Institute, Whittier, California
  - Memorial UC Health, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Research Institute, LLC., Plantation, Florida
  - Florida Cancer Specialists - North (FCS North), St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists - East (FCS East), West Palm Beach, Florida
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Community Health Network, Indianapolis, Indiana
  - University of Maryland Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - The University of Maryland St. Joseph Medical Center, Towson, Maryland
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Levine Cancer Center, Charlotte, North Carolina
  - Forsyth Memorial Hospital, Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Tennessee Oncology, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology-Dallas Presbyterian Hospital, Austin, Texas
  - Texas Oncology, P.A., Austin, Texas
  - Texas Oncology, P.A., Bedford, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-El Paso Cancer Treatment Center Grandview, El Paso, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Texas Oncology-San Antonio Northeast, San Antonio, Texas
  - Tyler Hematology-Oncology, PA, Tyler, Texas
  - Texas Oncology, P.A., Tyler, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Antwerp University Hospital (UZA), Edegem, Belgium
- Bulgaria (4):
  - University Multiprofile Hospital for Active Treatment, Sofia
  - MHAT for Womens Health - Nadezhda OOD, Sofia
  - Special Hospital For Active Treatment In Oncology, Sofia
  - Multiprofile Hospital for Active Treatment, Varna
- Croatia (4):
  - University Hospital Centre Osijek, Osijek
  - General Hospital Varaždin, Varaždin
  - University Hospital Centre "Sestre milosrdnice", Zagreb
  - University Hospital Centre Zagreb, Zagreb
- North Macedonia (2):
  - Clinical Hospital Dr. Trifun Panovski, Bitola
  - University Clinic of Radiotherapy and Oncology, Skopje
- Serbia (5):
  - Special Hospital for Internal Diseases , Oncomed, Belgrade
  - Clinical Hospital Centre Bezanijska Kosa, Oncology Clinic, Belgrade
  - Oncology Institute of Vojvodina, Clinic for Internal Oncology, Kamenitz
  - Center for Oncology and Radiotherapy, Clinical Centre, Kragujevac
  - Clinical Centre Nis, Clinic of Oncology, Niš
- Slovakia (2):
  - Mammacentrum, Sv.Agáty, Banská Bystrica
  - Cancer Institute VOU, Rastislavova, Košice
- University Medical Centre Maribor, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan AR, Wright GS, Thummala AR, Danso MA, Popovic L, Pluard TJ, Han HS, Vojnovic Z, Vasev N, Ma L, Richards DA, Wilks ST, Milenkovic D, Yang Z, Antal JM, Morris SR, O'Shaughnessy J. Trilaciclib plus chemotherapy versus chemotherapy alone in patients with metastatic triple-negative breast cancer: a multicentre, randomised, open-label, phase 2 trial. Lancet Oncol. 2019 Nov;20(11):1587-1601. doi: 10.1016/S1470-2045(19)30616-3. Epub 2019 Sep 28. PMID 31575503
- [Background] Tan AR, Wright GS, Thummala AR, Danso MA, Popovic L, Pluard TJ, Han HS, Vojnovic Z, Vasev N, Ma L, Richards DA, Wilks ST, Milenkovic D, Xiao J, Sorrentino J, Horton J, O'Shaughnessy J. Trilaciclib Prior to Chemotherapy in Patients with Metastatic Triple-Negative Breast Cancer: Final Efficacy and Subgroup Analysis from a Randomized Phase II Study. Clin Cancer Res. 2022 Feb 15;28(4):629-636. doi: 10.1158/1078-0432.CCR-21-2272. PMID 34887261

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 34 sites in the United States (US), Belgium, Bulgaria, Croatia, Republic of Macedonia, and Serbia from 02 February 2017 (first participant enrolled) to 28 February 2020 (last participant last visit).
Pre-assignment Details: Participants were screened within 28 days before the first dose of the treatment. Informed consent was obtained up to 28 days prior to first study drug administration. For tumor assessment, all sites of disease were assessed radiologically at screening. A total of 102 participants were randomized in this study.
Groups:
- Group 1: Gemcitabine/Carboplatin (Days 1 and 8): Participants received Intravenous (IV) infusion of standard GC chemotherapy (gemcitabine 1000 milligrams per meter square [mg/m^2] and carboplatin area under the curve [AUC] 2) on Days 1 and 8 of 21-day cycles. The carboplatin dose was calculated using the Calvert formula, with a target AUC 2 (maximum 300 mg).
- Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8): Participants received IV infusion of trilaciclib 240 mg/m^2 plus GC chemotherapy (gemcitabine 1000 mg/m^2 and carboplatin AUC 2) IV infusion on Days 1 and 8 of 21-day cycles. Trilaciclib was administered prior to chemotherapy.
- Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9): Participants received IV infusion of trilaciclib 240 mg/m^2 on Days 1, 2, 8, and 9 plus GC chemotherapy (gemcitabine 1000 mg/m^2 and carboplatin AUC 2) IV infusion on Day 2 and 9 of 21-day cycles. Trilaciclib was administered prior to chemotherapy.
Period: Overall Study
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Started | 34 | 33 | 35
ITT Population (The Intent-to-Treat (ITT) analysis set included all randomized participants.) | 34 | 33 | 35
Safety Analysis Set (The safety analysis set included all enrolled participants who received at least 1 dose of study drug.) | 30 | 33 | 35
Treated | 30 | 33 | 35
Completed | 0 | 0 | 0
Not Completed | 34 | 33 | 35
Not completed — Death | 25 | 13 | 20
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 6 | 4 | 5
Not completed — Sponsor terminated | 2 | 13 | 9
Not completed — Other | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The ITT analysis set included all randomized participants.
Groups:
- Group 1: Gemcitabine/Carboplatin (Days 1 and 8): Participants received IV infusion of standard GC chemotherapy (gemcitabine 1000 mg/m^2 and carboplatin AUC 2) on Days 1 and 8 of 21-day cycles. The carboplatin dose was calculated using the Calvert formula, with a target AUC 2 (maximum 300 mg).
- Total: Total of all reporting groups
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9) | Total
Number analyzed (Participants) | 34 | 33 | 35 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (13.6) | 56 (12.1) | 58 (9.5) | 56 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 35 | 101
  Male | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 2 | 9
  Not Hispanic or Latino | 32 | 28 | 33 | 93
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 7 | 2 | 14
  White | 28 | 22 | 28 | 78
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Duration of Severe (Grade 4) Neutropenia (DSN) During Cycle 1
Description: DSN was defined as the number of days from the date of the first absolute neutrophil count (ANC) value of less than (<) 0.5 × 10^9 cells/liter (L) observed between Day 1 Cycle 1 and the end of Cycle 1 to the date of the first ANC value greater than or equal to (>=) 0.5 × 10^9/L that met the following: (1) occurred after the ANC value of < 0.5 × 10^9 cells/L and (2) no other ANC values < 0.5 × 10^9 cells/L occurred between this day and the end of Cycle 1. Severe neutropenia (SN) was set to zero for participants who did not experience severe (Grade 4) neutropenia in Cycle 1, including those who were randomized but never treated.
Time Frame: From randomization to the end of Cycle 1 (Each cycle= 21 days)
Population: The ITT analysis set included all randomized participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 34 | 33 | 35
days | 1 (2.2) | 2 (3.5) | 1 (2.6)
Statistical Analysis 1: Comparison: Group 1: Gemcitabine/Carboplatin (Days 1 and 8) vs Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9); Duration of SN in Cycle 1 in Group 3 vs Group 1; Test type: Superiority; p = 0.7048, Analysis of covariance (ANCOVA) — A Hochberg-based gatekeeping procedure was used to control the global family-wise error rate across the multiple null hypotheses in the strong sense at a 1-sided 0.025 level; Mean difference = 0.3, 95% CI 2-sided [-0.8 to 1.5], Standard Error of Mean 0.58
Statistical Analysis 2: Comparison: Group 1: Gemcitabine/Carboplatin (Days 1 and 8) vs Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8); Duration of SN in Cycle 1 in Group 2 vs Group 1; Test type: Superiority; p = 0.3364, ANCOVA — 2-sided p-value was calculated using a ANCOVA with study baseline ANC value as covariate, stratification factors of lines of systemic therapy, liver involvement and treatment as fixed effects; Mean difference = 0.8, 95% CI 2-sided [-0.6 to 2.3], Standard Error of Mean 0.71

2. Primary Outcome: Number of Participants With Severe (Grade 4) Neutropenia (SN)
Description: Number of participants with Grade 4 SN was a binary variable. If a participants had at least 1 ANC value < 0.5 ×10^9/L during the treatment period, the participants was assigned as "yes" to the occurrence of SN. Otherwise, it was "no".
Time Frame: During the treatment period. From date of randomization, 21 day treatment cycles continue until disease progression, unacceptable toxicity, or discontinuation by the patient or investigator, assessed up to a maximum of 542 days
Population: The ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 34 | 33 | 35
Participants
  Grade 4 neutropenia: Yes | 9 | 12 | 8
  Grade 4 neutropenia: No | 25 | 21 | 27
Statistical Analysis 1: Comparison: Group 1: Gemcitabine/Carboplatin (Days 1 and 8) vs Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9); Number of participants with SN in Group 3 vs Group 1; Test type: Superiority; p = 0.7048, Modified Poisson method — A 1-sided p-value was calculated using Hochberg-based gatekeeping procedure to control the global familywise error rate across the multiple null hypotheses; Adjusted rate ratio = 0.776, 95% CI 2-sided [0.386 to 1.559], Standard Error of Mean 0.2762
Statistical Analysis 2: Comparison: Group 1: Gemcitabine/Carboplatin (Days 1 and 8) vs Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8); Number of participants with SN in Group 2 vs Group 1; Test type: Superiority; p = 0.9154, Modified Poisson Regression — The p-value was calculated using modified Poisson method adjusting for number of cycles, accounting for the number of prior lines of therapy (0 versus 1 - 2) and liver involvement as the stratification factors and baseline ANC as a covariate; Adjusted rate ratio = 0.961, 95% CI 2-sided [0.457 to 2.019], Standard Error of Mean 0.3640

3. Secondary Outcome: Number of Participants With Best Overall Response (BOR) as Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: BOR was defined as the best response across all time points (RECIST v1.1). The best overall response was determined once all the data for the participant is known. Each participant has been assigned one of the following categories (RECIST 1.1): complete response (CR): disappearance of all target lesions; partial response (PR): >= 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; progression disease (PD): >= 20% increase in the sum of diameters of target lesions (taking as reference the smallest sum on study); stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD); NE: not evaluable and missing.
Time Frame: From date of randomization until the occurrence of progressive disease or a censoring event, assessed up to a maximum of 875 days
Population: The response-evaluable (RE) analysis set included all participants who were in the modified intent-to-treat (mITT) analysis set, had measurable disease (target lesions [TLs]) at the baseline tumor assessment, and had (1) at least 1 post-baseline tumor assessment, (2) clinical progression (as noted by the investigator) before their first post-baseline tumor scan, or (3) died due to disease progression before their first post-baseline tumor scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 24 | 30 | 31
Participants
  Complete response (CR) | 0 | 0 | 0
  Partial response (PR) | 7 | 15 | 11
  Stable disease (SD) | 11 | 9 | 15
  Progressive disease (PD) | 6 | 5 | 3
  Not evaluable (NE) | 0 | 0 | 1
  Missing | 0 | 1 | 1

4. Secondary Outcome: Duration of Objective Response (DOR) as Per RECIST v1.1 as Determined by Investigator
Description: DOR is the time between first response by RECIST Version 1.1 of CR or PR and the first date that progressive disease is documented by RECIST Version 1.1, or death. Participants who do not experience PD or death was censored at the last tumor assessment date. 95% Confidence Interval (CI) was calculated using the Kaplan-Meier method.
Time Frame: as for outcome 3
Population: The RE analysis set included all participants who were in the mITT analysis set, had measurable disease TLs at the baseline tumor assessment, and had (1) at least 1 post-baseline tumor assessment, (2) clinical progression (as noted by the investigator) before their first post-baseline tumor scan, or (3) died due to disease progression before their first post-baseline tumor scan. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 7 | 15 | 11
months | 7.8 [7.5 to NA] — Due to small number of events, estimates (upper limit of 95% Confidence interval) from Kaplan-Meier survival curves could not be derived. | 11.5 [4.8 to 17.8] | 9.6 [3.1 to 12.6]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time (months) from date of randomization to the date of death due to any cause. Participants who do not die during the study were censored at the date last known to be alive. The OS was calculated using Kaplan-Meier method.
Time Frame: From date of randomization to date of death due to any cause, assessed up to a maximum of 1120 days
Population: The ITT analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 34 | 33 | 35
months | 12.6 [6.3 to 15.6] | NA [10.2 to NA] — Data could not be estimated due to higher number (>50%) of censored participants. | 17.8 [12.9 to 32.7]
Statistical Analysis 1: Comparison: Group 1: Gemcitabine/Carboplatin (Days 1 and 8) vs Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9); Overall survival in Group 3 vs Group 1; Test type: Superiority; p = 0.0004, stratified log-rank test — P-value was calculated using the stratified log-rank test to account for the number of prior lines of therapy (0 versus 1 - 2) and liver involvement as the stratification factors; Adjusted hazard ratio (HR) = 0.40, 95% CI 2-sided [0.22 to 0.74], Standard Error of Mean 0.125 — Cox regression model
Statistical Analysis 2: Comparison: Group 1: Gemcitabine/Carboplatin (Days 1 and 8) vs Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8); Overall survival in Group 2 vs Group 1; Test type: Superiority; p = 0.0016, stratified log-rank test — [p-value comment as in outcome 5, analysis 1]; Adjusted HR = 0.31, 95% CI 2-sided [0.15 to 0.63], Standard Error of Mean 0.111 — Cox regression model

6. Secondary Outcome: Progression Free Survival (PFS) as Per RECIST v1.1 as Determined by Investigator
Description: PFS was defined as the time (months) from date of randomization until date of documented PD or death due to any cause, whichever comes first. PD: >= 20% increase in the sum of diameters of target lesions (taking as reference the smallest sum on study). The PFS was calculated using Kaplan-Meier method.
Time Frame: From date of randomization until the occurrence of disease progression, death due to any cause or a censoring event, assessed up to a maximum of 875 days
Population: The ITT analysis set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 34 | 33 | 35
months | 5.7 [3.3 to 9.2] | 9.4 [6.1 to 11.9] | 7.3 [6.2 to 13.9]

7. Secondary Outcome: Relative Dose Intensity of Gemcitabine and Carboplatin
Description: Relative dose intensity was defined as 100% times the actual dose intensity divided by the planned dose intensity. The planned dose intensity was defined as the cumulative planned dose through the study divided by (number of cycles × 3 weeks). Relative dose intensity (%) was calculated as: for gemcitabine (100 * [Dose intensity (mg/m2/week) / (2000/3 (mg/m2/week)]); for carboplatin (100 * [Dose intensity (AUC/week)/ (4/3) (AUC/week)]) and for trilaciclib (100 * [Dose intensity (mg/m2/week)/ (480 /3 (mg/m2/week)] for Group 2 and 100 * [Dose intensity (mg/m2/week) / (960 /3 (mg/m2/week)] for Group 3).
Time Frame: During the treatment period. From date of first dose, 21 day treatment cycles continue until disease progression, unacceptable toxicity, or discontinuation by the patient or investigator, assessed up to a maximum of 871 days
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 30 | 33 | 35
percentage of dose
  Carboplatin | 77.5 (19.20) | 79.1 (15.88) | 81.7 (16.09)
  Gemcitabine | 79.1 (18.29) | 80.8 (12.51) | 81.0 (14.49)

8. Secondary Outcome: Duration of Exposure
Description: Duration of exposure (days) = First dose date of study drug from the last cycle - first dose date of study drug + 21.
Time Frame: as for outcome 7
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: days
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 30 | 33 | 35
days | 101 [21 to 469] | 161 [42 to 637] | 168 [21 to 436]

9. Secondary Outcome: Number of Cycles Participants Received Treatment in Each Treatment Arm
Description: Participants were considered to have started a cycle if they have received at least 1 dose of any study drug.
Time Frame: as for outcome 7
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: number of cycles
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 30 | 33 | 35
number of cycles | 6 (5.0) | 9 (6.6) | 8 (4.8)

10. Secondary Outcome: Cumulative Dose of Gemcitabine
Description: Cumulative dose: Sum of the total doses by cycle administered to a participant in the duration of exposure, i.e. total number of cycles received (milligram per meter square [mg/m^2]).
Time Frame: as for outcome 7
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/m^2
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 30 | 33 | 35
mg/m^2 | 10694.3 (9029.11) | 14680.9 (11557.90) | 13277.2 (8722.51)

11. Secondary Outcome: Cumulative Dose of Carboplatin
Description: Cumulative dose: Sum of the total doses by cycle (AUC) administered to a participant in the duration of exposure, i.e. total number of cycles received (in total prescribed AUC).
Time Frame: as for outcome 7
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: AUC (mg/mL/min)
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 30 | 33 | 35
AUC (mg/mL/min) | 20.3 (16.47) | 27.8 (21.21) | 26.0 (16.33)

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Trilaciclib
Description: The observed peak plasma concentration was determined from the plasma concentration-versus time data.
Time Frame: Cycle 1 Day 1 (Group 1): Pre-dose, 0.5, 1, 2, 3.5, 5, 24 hours post-dose; Cycle 1 Day 1 (Group 2) and Cycle 1 Day 2 (Group 3): Pre-dose, 0.5, 1, 1.5, 2.5, 4, 5.5, 24 hours post-dose (Each cycle is of 21 days)
Population: The pharmacokinetic (PK) analysis set included all dosed participants with evaluable PK data. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. Since, no participant received Trilaciclib in Group 1, data was not assessed and reported.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Group 1: Gemcitabine/Carboplatin (Day 1 and 8): Participants received IV infusion of standard GC chemotherapy (gemcitabine 1000 mg/m^2 and carboplatin AUC 2) on Days 1 and 8 of 21-day cycles. The carboplatin dose was calculated using the Calvert formula, with a target AUC 2 (maximum 300 mg).
Arm/Group | Group 1: Gemcitabine/Carboplatin (Day 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 0 | 6 | 7
ng/mL |  | 2280 (1790) | 1630 (423)

13. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to t Hours (AUC0-t) of Trilaciclib
Description: AUC0-t was calculated with the linear/log-trapezoidal method, which uses linear interpolation between data points to calculate the AUC. The linear/log-trapezoidal method will be employed for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from decreasing concentrations.
Time Frame: as for outcome 12
Population: The PK analysis set included all dosed participants with evaluable PK data. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. Since, no participant received Trilaciclib in Group 1, data was not assessed and reported.
Measure: Mean (Standard Deviation); unit: hour* nanogram per milliliter (h*ng/mL)
Arm/Group | Group 1: Gemcitabine/Carboplatin (Day 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 0 | 6 | 7
hour* nanogram per milliliter (h*ng/mL) |  | 3610 (1870) | 3800 (910)

14. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of Trilaciclib
Description: t1/2 was calculated as 0.693 divided by lambda z. lambda z (terminal phase rate constant) was determined by linear regression of at least 3 points on the terminal phase of the log-linear plasma concentration-time curve, the actual body exposure to drug after administration of a dose of the drug ( in mg*h/L).
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1: Gemcitabine/Carboplatin (Day 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 0 | 5 | 6
hours |  | 5.27 [3.98 to 6.64] | 5.31 [4.36 to 6.29]

15. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Gemcitabine
Description: The observed peak plasma concentration was determined from the plasma concentration-versus time data.
Time Frame: as for outcome 12
Population: The PK analysis set included all dosed participants with evaluable PK data. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Group 1: Gemcitabine/Carboplatin (Day 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 1 | 5 | 5
microgram per milliliter (mcg/mL) | NA (NA) — Data was not available since only one participant had sample in Group 1 and it was sufficient only for assessment of carboplatin. | 18.0 (4.04) | 23.8 (25.9)

16. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to t Hours (AUC0-t) of Gemcitabine
Description: AUC0-t was calculated with the linear/log-trapezoidal method.
Time Frame: as for outcome 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: hour*microgram per milliliter (h*mcg/mL)
Arm/Group | Group 1: Gemcitabine/Carboplatin (Day 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 1 | 5 | 5
hour*microgram per milliliter (h*mcg/mL) | NA — Data was not available since only one participant had sample in Group 1 and it was sufficient only for assessment of carboplatin. | 20.4 (11.6) | 15.4 (7.11)

17. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of Free Carboplatin
Description: t1/2 was calculated as 0.693 divided by lambda z. lambda z (terminal phase rate constant) was determined by linear regression of at least 3 points on the terminal phase of the log-linear plasma concentration-time curve.
Time Frame: as for outcome 12
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 1 | 5 | 5
hours | 5.23 | 2.49 [1.32 to 2.93] | 1.79 [1.35 to 4.86]

18. Secondary Outcome: Clearance (CL) of of Free Carboplatin
Description: Clearance after intravenous infusion administration was calculated as: CL=Dose/AUC0-inf. AUC0-inf was calculated as: AUC0-inf=AUClast+Clast/lambdaz where Clast is the last quantifiable concentration in the terminal elimination phase.
Time Frame: as for outcome 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Liter/hour (L/h)
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 1 | 3 | 5
Liter/hour (L/h) | 6.65 | 14.0 (2.80) | 13.7 (4.48)

19. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Free Carboplatin
Description: Vss was the volume of distribution at steady state of free carboplatin was reported.
Time Frame: as for outcome 12
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 1 | 5 | 5
Liter | 44.4 | 35.0 (12.0) | 34.0 (8.99)

20. Secondary Outcome: Number of Participants With Grade 3 and 4 Hematologic Toxicities
Description: Hematologic toxicities events were defined as any cycle where any hematologic lab value occurs that meets the CTCAE toxicity grade criteria for >= Grade 3 and the value is treatment emergent. The occurrence of Grade 3 and 4 hematologic toxicities was a binary endpoint. If a participant had at least 1 cycle with at least one Grade 3 or 4 hematologic toxicities during the treatment period, the participant was assigned as Yes to the occurrence of Grade 3 and 4 hematologic toxicities; otherwise, it was No. If a participant did not have an event, the value of 0 was assigned to that participant.
Time Frame: as for outcome 2
Population: The ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 34 | 33 | 35
Participants
  Participants with Grade 3 and 4 hematologic toxicities: Yes | 25 | 30 | 27
  Participants with Grade 3 and 4 hematologic toxicities: No | 9 | 3 | 8

21. Secondary Outcome: Number of Participants With Grade 3 or 4 Thrombocytopenia
Description: Hematologic toxicities events are defined as any cycle where any hematologic lab value occurs that meets the CTCAE toxicity grade criteria for >= Grade 3 and the value is treatment emergent. The occurrence of Grade 3 and 4 thrombocytopenia was a binary endpoint. If a participant had at least 1 cycle with at least one Grade 3 or 4 thrombocytopenia during the treatment period, the participant was assigned as "Yes" to the occurrence of Grade 3 and 4 thrombocytopenia; otherwise, it was "No". If a participant did not have an event, the value of 0 was assigned to that participant.
Time Frame: as for outcome 2
Population: The ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 34 | 33 | 35
Participants | 21 | 12 | 19

22. Secondary Outcome: Major Adverse Hematologic Event (MAHE) Rate
Description: MAHE was a composite endpoint incorporating the measurement of several clinically meaningful aspects of myelosuppression into a single endpoint by summing of the total number of events across a set of pre-specified components.The individual components for MAHE were all-cause hospitalizations, all-cause dose reductions, febrile neutropenia, prolonged severe neutropenia (duration > 5 days), RBC transfusion and platelet transfusion. Event rate for MAHE was calculated as the number of events/durations of treatment period divided by 7 days/1 week.
Time Frame: as for outcome 2
Population: The ITT analysis set included all randomized participants.
Measure: Number; unit: event rate per week
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 34 | 33 | 35
event rate per week | 0.153 | 0.108 | 0.080

23. Secondary Outcome: Number of Participants With Febrile Neutropenia (FN)
Description: The criterion for identifying FN was if the PT was "FEBRILE NEUTROPENIA" the occurrence during the treatment period was defined as a binary variable (Yes or No); Yes if total number of events >=1 was observed, No for other scenarios. If a participant did not have an event, the value of 0 was assigned to that participant.
Time Frame: as for outcome 2
Population: The ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 34 | 33 | 35
Participants | 1 | 1 | 0

24. Secondary Outcome: Number of Participants With Infection SAEs
Description: Number of participants with infection SAEs during the treatment period was defined as a binary variable (Yes or No); Yes if total number of events >=1 was observed, No for other scenarios. If a participant did not have an event, the value of 0 was assigned to that participant. The criterion for identifying the proper infection SAE records was as follows: If the system organ class (SOC) from Medical Dictionary for Regulatory Activities (MedDRA) takes value "INFECTIONS AND INFESTATIONS," and the AE was a serious event.
Time Frame: as for outcome 2
Population: The ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 34 | 33 | 35
Participants
  Participants with Infection SAEs: Yes | 2 | 0 | 0
  Participants with Infection SAEs: No | 32 | 33 | 35

25. Secondary Outcome: Number of Participants With Red Blood Cell (RBC) Transfusions On/After Week 5 (Day 35)
Description: Each RBC transfusion with a unique start date on/after 5 weeks on study during the treatment period was defined as a separate event. Occurrence during the treatment period was defined as a binary variable (Yes or No); "Yes" if the total number of events >=1 was observed and "No" for other scenarios. If a participant did not have an event, the value of 0 will be assigned to that participant.
Time Frame: From Day 35 through the treatment period. From date of randomization, 21 day treatment cycles continue until disease progression, unacceptable toxicity, or discontinuation by the patient or investigator, assessed up to a maximum of 508 days
Population: The ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 34 | 33 | 35
Participants
  Participants with RBC transfusions on/after Week 5: Yes | 12 | 11 | 8
  Participants with RBC transfusions on/after Week 5: No | 22 | 22 | 27
Statistical Analysis 1: Comparison: Group 1: Gemcitabine/Carboplatin (Days 1 and 8) vs Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9); RBC Transfusions in Group 3 vs Group 1; Test type: Superiority; p = 0.7048, modified Poisson regression — [p-value comment as in outcome 2, analysis 1]; Adjusted HR = 0.493, 95% CI 2-sided [0.226 to 1.073], Standard Error of Mean 0.1957
Statistical Analysis 2: Comparison: Group 1: Gemcitabine/Carboplatin (Days 1 and 8) vs Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8); RBC Transfusions in Group 2 vs Group 1; Test type: Superiority; p = 0.7272, Modified Poisson Regression — P-value was calculated using modified Poisson method adjusting for duration of treatment in days accounting for number of prior lines of therapy (0 versus 1 - 2); liver involvement as the stratification factors and baseline hemoglobin as a covariate; Adjusted rate ratio = 0.885, 95% CI 2-sided [0.447 to 1.754], Standard Error of Mean 0.3089

26. Secondary Outcome: Number of Participants With Platelet Transfusions
Description: Each platelet transfusion with a unique start date during the treatment period was defined as a separate event. The occurrence during the treatment period was defined as a binary variable (Yes or No); Yes if the total number of events >=1 was observed and No for other scenarios. If a participant did not have an event, the value of 0 will be assigned to that participant.
Time Frame: as for outcome 2
Population: The ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 34 | 33 | 35
Participants
  Participants with platelet transfusion: Yes | 4 | 3 | 6
  Participants with platelet transfusion: No | 30 | 30 | 29
Statistical Analysis 1: Comparison: Group 1: Gemcitabine/Carboplatin (Days 1 and 8) vs Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9); Platelet Transfusions in Group 3 vs Group 1; Test type: Superiority; p = 0.7048, modified Poisson regression — [p-value comment as in outcome 2, analysis 1]; Adjusted rate ratio = 0.988, 95% CI 2-sided [0.294 to 3.317], Standard Error of Mean 0.6105
Statistical Analysis 2: Comparison: Group 1: Gemcitabine/Carboplatin (Days 1 and 8) vs Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8); Platelet Transfusions in Group 2 vs Group 1; Test type: Superiority; p = 0.4078, Modified Poisson Regression — P-value: calculated using modified Poisson method adjusting for duration of treatment in days accounting for number of prior lines of therapy (0 versus 1 - 2); liver involvement as stratification factors and baseline platelet count as a covariate; Adjusted rate ratio = 0.527, 95% CI 2-sided [0.116 to 2.399], Standard Error of Mean 0.4077

27. Secondary Outcome: Number of Participants With Granulocyte Colony-stimulating Factor (G-CSF) Administration
Description: The criterion for selecting proper records is as follows: If the chemical subgroup from the World Health Organization-Drug Dictionary (WHO-DD) takes value "COLONY STIMULATING FACTOR," the medication was classified as G-CSF. The occurrence during the treatment period was defined as a binary variable (Yes or No); "Yes" if the total number of events >=1 was observed and "No" for other scenarios. If a participant did not have an event, the value of 0 will be assigned to that participant.
Time Frame: as for outcome 2
Population: The ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 34 | 33 | 35
Participants
  Participants with G-CSF Administration: Yes | 16 | 21 | 14
  Participants with G-CSF Administration: No | 18 | 12 | 21
Statistical Analysis 1: Comparison: Group 1: Gemcitabine/Carboplatin (Days 1 and 8) vs Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9); G-CSF Administration in Group 3 vs Group 1; Test type: Superiority; p = 0.7048, modified Poisson regression — [p-value comment as in outcome 2, analysis 1]; Adjusted rate ratio = 0.645, 95% CI 2-sided [0.362 to 1.150], Standard Error of Mean 0.1902
Statistical Analysis 2: Comparison: Group 1: Gemcitabine/Carboplatin (Days 1 and 8) vs Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8); G-CSF Administration in Group 2 vs Group 1; Test type: Superiority; p = 0.7835, Modified Poisson Regression — P-value was calculated using modified Poisson method adjusting for number of cycles, accounting for the number of prior lines of therapy (0 versus 1 - 2) and liver involvement as the stratification factors and baseline ANC as a covariate; Adjusted rate ratio = 0.936, 95% CI 2-sided [0.583 to 1.502], Standard Error of Mean 0.2260

28. Secondary Outcome: Number of Participants With Erythropoiesis Stimulating Agent (ESA) Administration
Description: The occurrence during the treatment period was defined as a binary variable (Yes or No); "Yes" if total number of events >=1 was observed, "No" for other scenarios. If a participant did not have an event, the value of 0 was assigned to that participant. The criterion to select proper records was as follows: If the chemical subgroup from WHO-DD Version September 2017 (i.e., TEXT4 for CODE4) takes value "OTHER ANTIANEMIC PREPARATIONS", the medication was classified as ESAs.
Time Frame: as for outcome 2
Population: The ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 34 | 33 | 35
Participants
  Participants with ESA Administration: Yes | 4 | 2 | 3
  Participants with ESA Administration: No | 30 | 31 | 32

29. Secondary Outcome: Number of Participants With Intravenous Antibiotics Use
Description: The criteria for identifying an IV antibiotic administration event was (1) if the Therapeutic subgroup from WHO-DD version takes value "ANTIBACTERIALS FOR SYSTEMIC USE", and (2) the route of medication was "intravenous" or the route was "other" with the detailed specification as "IVPB". The occurrence during the treatment period was defined as a binary variable (Yes or No); "Yes" if total number of events >=1 was observed, "No" for other scenarios. If a participant did not have an event, the value of 0 was assigned to that participant.
Time Frame: as for outcome 2
Population: The ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Day 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 34 | 33 | 35
Participants
  Participants with Intravenous Antibiotics Use: Yes | 6 | 5 | 0
  Participants with Intravenous Antibiotics Use: No | 28 | 28 | 35

30. Secondary Outcome: All-cause Dose Reductions, Event Rate (Per Cycle)
Description: Dose reductions were not permitted for trilaciclib. Dose reductions for gemcitabine or carboplatin were collected on the dosing page. No more than 3 dose modifications for toxicity in total were allowed for any participant. All dose reductions were counted as a separate event. Discontinuations of an individual component of the chemotherapy regimen were counted as a dose reduction If the participant continued the other chemotherapy drug as a monotherapy. Event rate was calculated as the total number of cycles with an event divided by the total number of cycles.
Time Frame: as for outcome 2
Population: The ITT analysis set included all randomized participants.
Measure: Number; unit: event rate per cycle
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 34 | 33 | 35
event rate per cycle | 0.141 | 0.118 | 0.133
Statistical Analysis 1: Comparison: Group 1: Gemcitabine/Carboplatin (Days 1 and 8) vs Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9); All-cause Dose Reductions in Group 3 vs Group 1; Test type: Superiority; p = 0.7048, negative binomial regression — The 1-sided p-value was calculated using Hochberg-based gatekeeping procedure to control the global family wise error rate across the multiple null hypotheses; Adjusted rate ratio = 0.991, 95% CI 2-sided [0.475 to 2.067], Standard Error of Mean 0.3718
Statistical Analysis 2: Comparison: Group 1: Gemcitabine/Carboplatin (Days 1 and 8) vs Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8); All-cause Dose Reductions in Group 2 vs Group 1; Test type: Superiority; p = 0.5541, negative binomial regression — P-value was calculated using negative binomial method adjusting for number of cycles, accounting for the number of prior lines of therapy (0 versus 1 - 2) and liver involvement as the stratification factors; Adjusted rate ratio = 0.820, 95% CI 2-sided [0.426 to 1.580], Standard Error of Mean 0.2744

31. Secondary Outcome: Dose Modifications: Number of Participants With Cycle Delays
Description: Dose modifications was summarized for each study drug based on number of cycles received during the treatment period. If the participant was unable to start a new cycle at that next visit, then the cycle is delayed, the reason entered, and the question was asked again at the next visit until the participant either starts a new cycle or discontinues treatment.
Time Frame: as for outcome 7
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 30 | 33 | 35
Participants | 17 | 19 | 22

32. Secondary Outcome: Dose Modifications - Number of Participants With Skipped Doses
Description: Dose modifications was summarized for each study drug based on skipped doses not received during the treatment period. Primary reasons for skipped doses included toxicity, investigator decision and administrative reasons (e.g., holidays).
Time Frame: as for outcome 7
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 30 | 33 | 35
Participants | 15 | 20 | 13

33. Secondary Outcome: Dose Modifications: Number of Participants With Any Dose Interruptions
Description: Dose interruptions was defined as interruption of infusion, regardless of whether the study drug was continued after the interruption.
Time Frame: as for outcome 7
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 30 | 33 | 35
Participants
  Trilaciclib | NA — Here, 'NA' signifies that Trilaciclib drug was not administered in this specified arm. | 3 | 5
  Carboplatin | 1 | 1 | 0
  Gemcitabine | 2 | 4 | 0

34. Secondary Outcome: Dose Modifications - Number of Participants With Dose Reductions
Description: Dose (mg/m2) reductions were not permitted for trilaciclib. Dose reductions for carboplatin and gemcitabine were determined by comparing the planned dose on the respective drug administration pages between the current cycle and the previous cycle.
Time Frame: as for outcome 7
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 30 | 33 | 35
Participants
  Carboplatin | 10 | 13 | 15
  Gemcitabine | 13 | 20 | 17

35. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An Adverse event (AE) was any untoward medical occurrence in a participant administered a medicinal product that did not necessarily have a causal relationship with this treatment. Any AE that started on or after the first dose of study drugs was included as a TEAE. A Serious AE was defined as any AE, occurring at any dose (including after the informed consent form was signed and prior to dosing) and regardless of causality that met one, more of the following criteria: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event. TEAEs included serious and non-serious TEAEs.
Time Frame: During the treatment period. From date of first dose, 21 day treatment cycles continue until disease progression, unacceptable toxicity, or discontinuation by the patient or investigator, assessed up to a maximum of 1116 days
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib + Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
Number analyzed (Participants) | 30 | 33 | 35
Participants
  Participants with any TEAEs | 30 | 33 | 34
  Participants with any Serious TEAEs | 10 | 11 | 4

ADVERSE EVENTS:
Time Frame: From date of randomization up to 1121 days
Description: Safety evaluations were conducted at baseline and throughout the study. Safety surveillance reporting of AEs and SAEs commenced at the time of informed consent and continued through 30 days after the last dose of study drug (safety follow-up phone call). The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Group 2: Trilaciclib (G1T28)+ Gemcitabine/Carboplatin (Days 1 and 8): Participants received IV infusion of trilaciclib 240 mg/m^2 plus GC chemotherapy (gemcitabine 1000 mg/m^2 and carboplatin AUC 2) IV infusion on Days 1 and 8 of 21-day cycles. Trilaciclib was administered prior to chemotherapy.
Arm/Group | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) | Group 2: Trilaciclib (G1T28)+ Gemcitabine/Carboplatin (Days 1 and 8) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9)
All-Cause Mortality (participants affected / at risk) | 25/30 | 13/33 | 20/35
Serious Adverse Events (participants affected / at risk) | 10/30 | 11/33 | 4/35
Other Adverse Events (participants affected / at risk) | 30/30 | 33/33 | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) (N=30) | Group 2: Trilaciclib (G1T28)+ Gemcitabine/Carboplatin (Days 1 and 8) (N=33) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9) (N=35)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Gemcitabine/Carboplatin (Days 1 and 8) (N=30) | Group 2: Trilaciclib (G1T28)+ Gemcitabine/Carboplatin (Days 1 and 8) (N=33) | Group 3: Trilaciclib (Days 1, 2, 8 and 9) + Gemcitabine/Carboplatin (Days 2 and 9) (N=35)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 1 (7)
Hot flush (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 3 (7)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 11 (17) | 14 (22) | 16 (35)
Oedema peripheral (General disorders) | 4 (5) | 4 (7) | 4 (8)
Pyrexia (General disorders) | 3 (3) | 6 (8) | 2 (2)
Pain (General disorders) | 5 (7) | 2 (2) | 3 (3)
Chills (General disorders) | 0 (0) | 6 (7) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 4 (5)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 2 (2)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 2 (4)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Mucosal inflammation (General disorders) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2) | 4 (4)
Depression (Psychiatric disorders) | 3 (3) | 5 (5) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1) | 4 (4)
Breast pain (Reproductive system and breast disorders) | 3 (3) | 1 (4) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 7 (35) | 4 (6)
Neutrophil count decreased (Investigations) | 8 (20) | 12 (50) | 11 (30)
Platelet count decreased (Investigations) | 8 (38) | 8 (13) | 12 (44)
Alanine aminotransferase increased (Investigations) | 3 (5) | 4 (6) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 3 (6) | 4 (5) | 4 (7)
White blood cell count decreased (Investigations) | 2 (7) | 4 (7) | 2 (5)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (3) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 22 (61) | 16 (46) | 15 (35)
Neutropenia (Blood and lymphatic system disorders) | 13 (49) | 15 (79) | 12 (31)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (68) | 13 (55) | 11 (55)
Leukopenia (Blood and lymphatic system disorders) | 5 (9) | 3 (12) | 1 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (10) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (8) | 7 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 6 (9) | 9 (11) | 14 (22)
Dizziness (Nervous system disorders) | 6 (8) | 4 (7) | 6 (11)
Dysgeusia (Nervous system disorders) | 0 (0) | 5 (5) | 1 (1)
Cognitive disorders (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (8) | 14 (19) | 17 (31)
Vomiting (Gastrointestinal disorders) | 8 (9) | 8 (23) | 11 (18)
Constipation (Gastrointestinal disorders) | 5 (6) | 9 (16) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 9 (15) | 5 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 5 (5) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 4 (6) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 2 (5) | 1 (1) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (4) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 4 (5)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (21) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (4) | 2 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (15) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (7) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (6) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (6) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (5) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 5 (6) | 4 (7)
Hypophosphataemia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 3 (7)
Dehydration (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (3) | 2 (2) | 2 (2)
Hypoalbuminaemia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 2 (2)
Hypocalcaemia (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (2) | 0 (0)
Hyperlipidaemia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 4 (4) | 3 (4)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations of this study are the small sample size and open-label design. Antitumor outcomes were not the primary endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator will submit results communications for review by the sponsor at least 60 days prior to expected submission to the intended publisher or meeting committee. This review period may be shortened upon mutual consent. The sponsor may request modification of any publication, presentation or use by the investigator if such activity may jeopardize a patent application, an existing patent, or other proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT02978716/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT02978716/SAP_001.pdf